CLINICAL TRIAL: NCT03015558
Title: Transcranial Direct Current Stimulation (tDCS) for Neuropathic Chronic Pain : Study of the Opercular-insular Cortex Stimulation
Brief Title: Analgesic Effect of Non Invasive Stimulation : Transcranial Direct Current Stimulation of Opercular-insular Cortex
Acronym: STIM-INSULA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 69HCL15_0345; 2016-A00022-49 (Other: ID-RCB)
Record Dates: First submitted 2016-12-22; First posted 2017-01-10 (Estimated); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Neuropathic Pain
Keywords: Drug Resistance; Neuropathic Pain; opercular-insular cortex; Transcranial Direct Current Stimulation
MeSH Terms: conditions — Neuralgia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- patients (Experimental)
  Interventions: Device: transcranial direct current stimulation of opercular-insular cortex - anodal active tDCS session; Device: transcranial direct current stimulation of opercular-insular cortex - active control session; Device: transcranial direct current stimulation of opercular-insular cortex - sham control session.
- healthy subjects (Active Comparator)
  Interventions: Device: transcranial direct current stimulation of opercular-insular cortex - anodal active tDCS session; Device: transcranial direct current stimulation of opercular-insular cortex - active control session; Device: transcranial direct current stimulation of opercular-insular cortex - sham control session.

INTERVENTIONS:
Device: transcranial direct current stimulation of opercular-insular cortex - anodal active tDCS session — transcranial direct current stimulations of opercular-insular cortex. Three sessions separated by a minimum of 2 weeks, with three different conditions: one session with anodal active tDCS, one with active control, and one with sham control.
Device: transcranial direct current stimulation of opercular-insular cortex - active control session — transcranial direct current stimulations of opercular-insular cortex. Three sessions separated by a minimum of 2 weeks, with three different conditions: one session with anodal active tDCS, one with active control, and one with sham control.
Device: transcranial direct current stimulation of opercular-insular cortex - sham control session. — transcranial direct current stimulations of opercular-insular cortex. Three sessions separated by a minimum of 2 weeks, with three different conditions: one session with anodal active tDCS, one with active control, and one with sham control.

SUMMARY:
The aim of this study is to evaluate, versus placebo, the analgesic efficacy of the opercular-insular cortex stimulation with Transcranial Direct Current Stimulation (tDCS), in both healthy subjects and chronic neuropathic pain patients. In healthy subjects analgesia by tDCS will be assessed using both laser stimuli and cold pressor test. In patients the assessment regards their chronic pain (ratings for ongoing, evoked and paroxysmal pain, sleep and fatigue). Opercular-insular stimulation is obtained via a combined 6-electrode montage and by bi-vestibular stimulation (since vestibular pathways reach the posterior insular cortex). In patients, three separate conditions (two active and one sham) will be tested in randomised order. In healthy subjects, two other conditions are added to control for attention and distraction confounders.

ELIGIBILITY:
Inclusion Criteria:

* healthy subjects aged from 18 to 70 years, male or female, with social security protection, fully informed and having given their written consent.
* patients aged from 18 to 80 years, male or female, with social security protection , fully informed and having given their written consent.
* pharmacoresistant neuropathic pain during at least one year,
* without any change of the pharmacological treatment since at least one month

Exclusion Criteria:

In healthy subjects only:

* history of chronic pain
* analgesic medication within 24h before stimulation

For patients only: new analgesic treatment within 1 month before consent

for both:

* drug addiction, headache, epilepsy
* ferromagnetic intracranial device
* implanted stimulator
* recent neurosurgery and open wound of the scalp.
* absence of contraceptive method for women of childbearing age

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2016-11-02 (Actual); Primary Completion 2018-03-28 (Actual); Study Completion 2018-03-28 (Actual)

PRIMARY OUTCOMES:
In healthy subjects : Change in subjective pain and (when applicable) in cortical evoked potentials with pain scale | just before the tDCS session at Day 0
In patients : Changes in daily ratings of global pain | just before the tDCS session at Day 0
In healthy subjects : Change in subjective pain and (when applicable) in cortical evoked potentials | just after the tDCS session at Day 0
In patients : Changes in daily ratings of global pain | just after the tDCS session at Day 0
In patients : Changes in daily ratings of global pain | at week 1

SECONDARY OUTCOMES:
ongoing pain with pain scale | just before the tDCS session at Day 0
ongoing pain with pain scale | just after the tDCS session at Day 0
ongoing pain as assessed by daily ratings | during one week

CONTACTS AND LOCATIONS:
Overall Officials: Luis GARCIA-LARREA, MD, Principal Investigator — NeuroPain lab - CRNL (Inserm U1028 - UCBL)
Locations (1):
- Hospices Civils de Lyon - NeuroPain lab - CRNL, Bron, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hagiwara K, Perchet C, Frot M, Bastuji H, Garcia-Larrea L. Cortical modulation of nociception by galvanic vestibular stimulation: A potential clinical tool? Brain Stimul. 2020 Jan-Feb;13(1):60-68. doi: 10.1016/j.brs.2019.10.009. Epub 2019 Oct 12. PMID 31636023